CLINICAL TRIAL: NCT02677857
Title: Developing a Healthy Lifestyle in Breast Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment efforts were not effective.
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTKIRB-15-02602-FB
Record Dates: First submitted 2016-01-25; First posted 2016-02-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer; Sedentary Lifestyle
MeSH Terms: conditions — Breast Neoplasms; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded

ARMS (3):
- Lifestyle (Active Comparator): Participants will be educated on the relationship between MVPA and improved health outcomes, including weight management, and cancer survivorship. The goal will be to increase MVPA to > 40 min/day 5 times/wk As participants will be overweight/obese, inactive, and coming into the program with different levels of baseline fitness and time since last cancer treatment, participants will shape their MVPA to meet the targeted goals. Initially, participants will be encouraged to complete MVPA > 10 min/day 5 times/wk, and then progressively increase MVPA by 5 min/day every week until reaching the intervention goal (week 7 of the 12 week intervention). Participants will be encouraged to do brisk walking and be allowed to accumulate time spent being physically active by engaging in multiple short bouts (i.e., > 10 min in length). Any MVPA in bouts of > 10 min in length will be counted towards the MVPA goal. Participants will self-monitor their MVPA using the Polar® Loop tracking system.
  Interventions: Behavioral: Common intervention components for Lifestyle
- Lifestyle + SB (Active Comparator): Participants will receive everything that is described in Lifestyle. Additionally, they will be educated on the relationship between SB and weight management, and cancer survivorship risk. The goal will be to reduce sedentary time by > 2 hrs/day or > 14 hrs/wk. Participants will shape towards the goal. Baseline measures will be used as the starting point from where to calculate the 2 hrs/day reduction, providing participants with a total SB goal per day. For example, if baseline measures indicate that a participant has a mean daily SB amount of 9.75 hrs, the participant's SB goal will be 7.75 hrs/day. To achieve that goal, participants will reduce SB by 20 minutes a day, starting week 2, with a decrease of an additional 20 minutes/day occurring weekly until the SB goal is achieved (week 7 of the 12 week intervention. Participants will self-monitor their SB using the Polar® Loop tracking system.
  Interventions: Behavioral: Common intervention components for Lifestyle
- Newsletter (No Intervention): Participants in this condition will receive standard care and every month they will receive a newsletter that provides information and tips about healthy eating and activity behaviors. This newsletter will include information on myPlate,28 activity guidelines,29 reading food labels, healthy recipes, and seasonal activity suggestions.

INTERVENTIONS:
Behavioral: Common intervention components for Lifestyle — Participants in these conditions will receive standard care and one of the Lifestyle conditions. There are several components that will be identical for both Lifestyle conditions. These components include treatment structure, dietary goals, and cognitive behavioral strategies.
  Arms: Lifestyle; Lifestyle + SB

SUMMARY:
At this time, no study has examined the effect of a lifestyle intervention with a reduced Sedentary Behavior (SB) prescription on overall physical activity, weight loss, metabolic dysfunction, and inflammation in breast cancer survivors. Thus, in collaboration with University of Tennessee Medical Center's (UTMC) Cancer Institute, investigators propose to randomize 30 female breast cancer survivors (history of breast cancer stages I [> 1 cm], II, or III) with a body mass index (BMI) between 25 and 45 kg/m2 who are sedentary (engage in > 8 hours a day of SB) and inactive (engage in < 100 min/wk MVPA) to one of three, 3-month conditions:

1. lifestyle intervention (Lifestyle) (increase MVPA to > 200 min/wk);
2. lifestyle intervention with a reduced SB prescription (Lifestyle+SB) (increase MVPA to > 200 min/wk and reduce SB by 2 hrs/day); or
3. weight management education materials provided via mailed newsletter (Newsletter).

Lifestyle and Lifestyle+SB will receive a standard dietary (low-calorie [1200-1500 kcal/day], low-fat [<30% calories from fat]) prescription that emphasizes intake of fruits, vegetables, and whole grains, and a cognitive behavioral intervention to assist with meeting activity and diet goals. Dependent variables, measured at 0 and 3 months, include objectively measured SB, LPA, MVPA, and total activity via accelerometry; self-reported SB; percent weight loss; insulin and glucose, and leptin and C-reactive protein (CRP) (biomarkers of cancer prognosis that have been found to be positively related to SB and/or adiposity); diet; body composition; and fitness.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 yrs
2. BMI between 25 and 45 kg/m2
3. history of breast cancer (stages I [> 1 cm], II, or III) diagnosed within the previous 5 years
4. completion of initial therapies
5. engage in > 8 hours a day of SB
6. engage in < 100 min/wk MVPA.

Exclusion Criteria:

1. report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q)25 (The Health Screening Questionnaire will also be used to identify individuals with joint problems, prescription medication usage, or other medical conditions that could limit exercise, and these individuals will be required to obtain written physician consent to participate - the two questionnaires are found in questions 4-11 in the phone screen in Appendix B)
2. report being unable to walk for 2 blocks (1/4 mile) without stopping
3. report major psychiatric diseases or organic brain syndromes
4. report a serious medical condition in which weight loss is contraindicated
5. are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months
6. have had bariatric surgery or are planning to have bariatric surgery in the next 6 months
7. are participating in a program to increase physical activity and/or decrease sedentary time
8. intend to move outside of the metropolitan area within the time frame of the investigation
9. are pregnant, lactating, < 6 months post-partum, or plan to become pregnant during the investigation
10. are unwilling to attend sessions and/or unwilling to be randomized to any treatment condition;
11. do not own a smartphone that will run the app required for the Polar® Loop device;
12. are unwilling to use MyFitnessPal or the Polar® Loop device app for smartphones; or
13. have a metal allergy or are not able to wear anything on an upper arm (which would prevent the ability of participant to wear the SenseWear® armband from BodyMedia® used in the proposed study).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measures of activity by Armband | change from baseline to 12 weeks
  Participants will wear the SenseWear Armband (SWA) for data collection of time spent engaging in physical activity per day.
Weight | change from baseline to 12 weeks
  Weight will be assessed by an electronic scale.
Measures of diet | change from baseline to 12 weeks
  Diet will be assessed by 3-day food records (2 weekdays and 1 weekend day). Each record will be completed using the Nutrition Data System Software for Research (NDS-R) developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
Fitness (The 6 Minute Walk Test (6MWT)) | change from baseline to 12 weeks
  The 6 Minute Walk Test (6MWT) is well tolerated by participants who are obese. Participants will walk as quickly as possible, without jogging or running, around two cones placed 60 m apart for 6 min. The primary measure will be distance walked. The 6MWT has been significantly correlated to peak oxygen uptake (VO2) values from a cycle ergometer test (r = .73, p < 0.001). The 6MWT has been shown to measure enhanced physical performance beyond that which occurs from weight loss itself in participants with obesity. Standard safety protocols will be used for participants that Dr. Bell considers appropriate for testing.
Physical activity by Questionnaire | change from baseline to 12 weeks
  Participants will complete the Past-day Adults' Sedentary Time (PAST), a seven-item questionnaire that asks questions about sedentary behaviors that have occurred during the previous day.
Insulin | change from baseline to 12 weeks
  Blood samples will be obtained from over-night fasted participants who have not engaged in MVPA and analyzed at UTMC using standard procedures.
Glucose | change from baseline to 12 weeks
  Blood samples will be obtained from over-night fasted participants who have not engaged in MVPA and analyzed at UTMC using standard procedures.
Leptin | change from baseline to 12 weeks
  Blood samples will be obtained from over-night fasted participants who have not engaged in MVPA and analyzed at UTMC using standard procedures.
C-Reactive Protein | change from baseline to 12 weeks
  Blood samples will be obtained from over-night fasted participants who have not engaged in MVPA and analyzed at UTMC using standard procedures.
Height | baseline
  Height will be assessed using a stadiometer at baseline
BMI | change from baseline to 12 weeks
  BMI (kg/m2) will be calculated from height and weight measurements.
Waist circumference | change from baseline to 12 weeks
  waist measurement
Percent body fat | change from baseline to 12 weeks
  Percent body fat will be assessed by bioelectrical impedance analysis (BIA), using the foot to foot pressure contact electrode BIA technique (Tanita TBF-300A model) following standard protocol

SECONDARY OUTCOMES:
Completion of self-monitoring records | 12 weeks
  Number of weekly records of self-monitoring of diet and activity completed and turned in.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States